CLINICAL TRIAL: NCT06275035
Title: Memantine to Preserve Memory and Neurocognition Following Craniospinal Irradiation- A Randomised Controlled Trial (MEMENTO)
Brief Title: Evaluation of Memantine in the Preservation of Memory and Neurocognition Following CSI
Acronym: MEMENTO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr. Tejpal Gupta, Dr Tejpal Gupta, Professor, Department of Radiation Oncology, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4235
Record Dates: First submitted 2024-01-17; First posted 2024-02-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Neurocognitive Dysfunction
MeSH Terms: conditions — Cognition Disorders | interventions — Memantine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Participants in the experimental arm (memantine) will be started on memantine. The starting dose of memantine will be 5mg once daily at bedtime for 1 week, followed by 5mg twice daily for 1 week, and finally increased to the full dose of 10 mg twice daily for 6 months.
  Interventions: Drug: Memantine Oral Tablet
- Standard arm (No Intervention): Participants in the standard arm will continue the standard treatment as planned.

INTERVENTIONS:
Drug: Memantine Oral Tablet — Drug to preserve memory and neurocognitive dysfunction induced by radiation therapy
  Other Names: Memantine
  Arms: Experimental arm

SUMMARY:
The goal of this clinical trial is to evaluate the role of memantine in preservation of memory and neurocognition in patients undergoing craniospinal irradiation. Participants will be randomised into two arms and the interventional arm will receive memantine along with the standard treatment. Researchers will compare the neurocognitive tests of participants in both the arms to see if memantine leads to significant preservation of memory and cognition post radiation therapy.

DETAILED DESCRIPTION:
Craniospinal irradiation (CSI) involving radiation (RT) of brain and spine, along with tumor-bed boost with or without chemotherapy, is the current standard treatment for medulloblastoma and other primitive embryonal tumors of the central nervous system (CNS). The delayed side effects following CSI include memory loss, hearing and balance difficulties, hormonal imbalance, and secondary cancers. Decline in memory severely affects the quality of life in long term survivors of these diseases. Hence, various strategies are being tried to prevent it. Memantine has been proven to effectively prevent the memory decline induced by RT. It is FDA-approved for Alzheimer's disease and is widely used in the children for several developmental disorders. With this study, we are trying to investigate the role of memantine in patients receiving CSI to prevent memory decline.

After screening for the study, eligible patients will be randomly allocated (by computerised system) to one of the two arms that are described as follows. Patients in the experimental arm (memantine) will be started on memantine, starting dose of the same will be 5mg once daily at bedtime for 1 week, followed by 5mg twice daily for 1 week, and finally increased to the full dose of 10 mg twice daily for 6 months. Patients will continue on radiation and chemotherapy (when indicated) as per schedule. All patients in the study will undergo neurocognitive evaluation, the time points for which will be pre-radiation (baseline), 6 months post-RT, 1-year post-RT, and annually after that for 5 years from radiation. Following completion of RT or treatment, standard follow-up protocols will include a clinical examination 3 monthly for the first 2 years, followed by 6 monthly visits till 5 years post-RT. No additional risk is expected from the current study other than the common side effects of the standard treatment. Based on the results from the study, if primary endpoints are achieved, it will establish the role of memantine in preventing memory decline from CSI, which can be used as a standard treatment measure to help patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age at irradiation: 5 to 39 years
* Planned for CSI (with or without boost dose) with or without systemic chemotherapy
* Informed consent or assent taken
* Karnofsky Performance Status / Lansky Performance Status ≥ 60

Exclusion Criteria:

* Re-irradiation
* Prior exposure to memantine
* Inability to undergo Wechsler test

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive-deterioration-free survival at 2 years | 2 years
  Cognitive-deterioration-free survival at 2 years; defined by a drop of 5 points in any of Full Scale Intelligence Quotient (FSIQ), Verbal Intelligence Quotient (VIQ), or Performance Intelligence Quotient (PIQ) compared to baseline (pre-radiation) on Wechsler Adult Intelligence Scale (WAIS), and Wechsler Intelligence Scale for Children (WISC).

SECONDARY OUTCOMES:
Full-Scale Intelligence Quotient (FSIQ) in children | 7 years
  The slope of decline of FSIQ with time as measured using age-appropriate neurocognitive test battery for children (Wechsler Intelligence Scale for Children- WISC)
Overall survival (OS) | 7 years
  Comparison of survival outcomes in both the arms
Academic performance by scholastic performance and grades | 7 years
  Comparison of scholastic performance as graded in school examinations in pediatric participants in both arms
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of Memantine | 2 years
  Recording of any unexpected adverse drug reactions according to CTCAE v 5.0
Progression-Free Survival (PFS) | 7 years
  Comparison of progression-free survival time in both arms
Full-Scale Intelligence Quotient (FSIQ) in adults | 7 years
  The slope of decline of FSIQ with time as measured using age-appropriate neurocognitive test battery for adults (Wechsler Adult Intelligence Scale-WAIS)

OTHER OUTCOMES:
Full Scale Intelligence Quotient change in subgroups | 7 years
  Subgroup analysis of FSIQ slope. Subgroup stratification based on age, prior treatment of chemotherapy, dose of radiation received
Radiological features of cognitive decline on Magnetic Resonance Imaging | 7 years
  Fractional decline in volume of anatomical structures like hippocampus with radiation and correlation with FSIQ using Pearson correlation.
Neuroinflammatory markers correlation with neurocognitive decline and survival | 7 years
  Neuro-inflammatory markers in Cerebrospinal Fluid (CSF), blood and its correlation with Full-Scale Intelligence Quotient scores.
  List of markers to be measured:-
  * Inflammatory panel using ELISA: Interleukin(IL)- 6, IL-1, IL-4, IL-8, IL-10, IL-11, IL-12, Tumor Necrosis Factor- alpha, Interferon- gamma, Granulocyte macrophage colony-stimulating factor, Chitinase-3-like protein 1, Transforming Growth Factor- beta, C- reactive protein, Glial Fibrillary Acidic Protein, Ubiquitin, Carboxy- terminal hydrolase L1
  * Cell free Deoxyribo Nucleic Acid- using MagMax cell free DNA isolation kit
  * Circulating cancer cells using cell search circulating tumor cell kit

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data from the study will not be shared publicly but anonymized data can be made available upon reasonable request to the Principal Investigator

REFERENCES:
- [Background] Brown PD, Pugh S, Laack NN, Wefel JS, Khuntia D, Meyers C, Choucair A, Fox S, Suh JH, Roberge D, Kavadi V, Bentzen SM, Mehta MP, Watkins-Bruner D; Radiation Therapy Oncology Group (RTOG). Memantine for the prevention of cognitive dysfunction in patients receiving whole-brain radiotherapy: a randomized, double-blind, placebo-controlled trial. Neuro Oncol. 2013 Oct;15(10):1429-37. doi: 10.1093/neuonc/not114. Epub 2013 Aug 16. PMID 23956241
- [Background] Brown PD, Gondi V, Pugh S, Tome WA, Wefel JS, Armstrong TS, Bovi JA, Robinson C, Konski A, Khuntia D, Grosshans D, Benzinger TLS, Bruner D, Gilbert MR, Roberge D, Kundapur V, Devisetty K, Shah S, Usuki K, Anderson BM, Stea B, Yoon H, Li J, Laack NN, Kruser TJ, Chmura SJ, Shi W, Deshmukh S, Mehta MP, Kachnic LA; for NRG Oncology. Hippocampal Avoidance During Whole-Brain Radiotherapy Plus Memantine for Patients With Brain Metastases: Phase III Trial NRG Oncology CC001. J Clin Oncol. 2020 Apr 1;38(10):1019-1029. doi: 10.1200/JCO.19.02767. Epub 2020 Feb 14. PMID 32058845